CLINICAL TRIAL: NCT06376565
Title: Multilevel Health System Intervention to Increase Guideline-Concordant Surveillance Colonoscopy for High Risk Colon Polyps
Brief Title: Improving Colonoscopy Surveillance for Patients With High Risk Colon Polyps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-000647; NCI-2024-02090 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA271034 (NIH)
Record Dates: First submitted 2024-04-10; First posted 2024-04-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I(Multilevel intervention) (Experimental): Aim 1: Participants complete an interview over 20-30 minutes.
  Aim 2: Clinics have the automatic addition of HRN to the medical problem list and indication of surveillance interval is added to the health maintenance portion of the electronic health records (EHR). Clinics also call patients to schedule their colonoscopy. Providers receive reminders and pending orders for the colonoscopy in the electronic health record. Patients receive a reminder 6 months in advance via their patient portal and mail to schedule a colonoscopy, and also receive a phone call from the patient communication center.
  Interventions: Other: Communication Intervention; Other: Interview
- Arm II (Standard follow up) (Active Comparator): Patients receive care according to the clinics' usual care practices.
  Interventions: Other: Best Practice; Other: Interview

INTERVENTIONS:
Other: Best Practice — Receive standard care
  Other Names: standard of care; standard therapy
  Arms: Arm II (Standard follow up)
Other: Communication Intervention — Complete clinic EHR interventions
  Arms: Arm I(Multilevel intervention)
Other: Communication Intervention — Receive scheduling reminders
  Arms: Arm I(Multilevel intervention)
Other: Communication Intervention — Receive reminders and pending EHR orders
  Arms: Arm I(Multilevel intervention)
Other: Interview — Complete interview
  Arms: Arm I(Multilevel intervention)
Other: Interview — Ancillary studies
  Arms: Arm II (Standard follow up)

SUMMARY:
This clinical trial tests a multilevel intervention at the clinic, provider and patient levels, to improve colonoscopy surveillance in patients with high risk colon polyps. Colorectal cancer (CRC) is a common and deadly disease that is largely preventable through the detection and removal of colorectal polyps. One million Americans are diagnosed with high risk polyps of the colon or rectum annually and are at increased risk for CRC; however, uptake of recommended repeat colonoscopy in 3 years to reduce CRC risk is low in this group. This multilevel intervention may work to improve timely colonoscopy screening for patients with high risk colon polyps.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To increase completion of surveillance colonoscopy within 3.5 years of high risk neoplasia (HRN) diagnosis.

OUTLINE:

AIM 1: Participants complete an interview over 20-30 minutes.

AIM 2: Primary care clinics are randomized to 1 of 2 arms.

ARM I: Clinics have the automatic addition of HRN to the medical problem list and indication of surveillance interval is added to the health maintenance portion of the electronic health records. Clinics also call patients to schedule their colonoscopy. Providers receive reminders and pending orders for the colonoscopy in the electronic health record. Patients receive a reminder 6 months in advance via their patient portal and mail to schedule a colonoscopy, and also receive a phone call from the patient communication center.

ARM II: Patients receive care according to the clinics' usual care practices.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 PATIENTS: Patients between age 45 and 75 with a HRN diagnosis in the past 5 years
* AIM 1 PATIENTS: 12 patients who did and 12 patients who did not have surveillance colonoscopy
* AIM 1 PROVIDERS: Primary care providers (PCPs) and gastroenterologists (GIs)
* AIM 1 ADMINISTRATORS: Administrators who are involved in care processes related to CRC screening, HRN surveillance, and/or colonoscopy scheduling
* AIM 2: Patients age 45 to 75 diagnosed with a HRN during the pre-specified two-year HRN diagnosis period

Exclusion Criteria:

* AIM 2: Individuals with a personal history of colorectal carcinoma (CRC), inflammatory bowel disease (Crohn's, ulcerative colitis), or polyposis syndrome
* AIM 2: HRN cases not confirmed by chart review (human-in-the-loop)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1680 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Stakeholder perspectives on the multilevel intervention (Aim 1) | At time of interview
  The Investigators will conduct 1-on-1 in-depth interviews with patients, advocates, providers, and administrators. these interviews will provide data in closer proximity to intervention implementation to optimize composition, timing, and acceptability of each component. Interview content is guided by the multiple health outcomes framework (MHOF) and addresses major barriers (patient, provider, system) to surveillance and challenges (patient, provider, system) to the planned implementation of intervention components.
Completion of surveillance colonoscopy (Aim 2) | At 3.5 years
  Will analyze rates during the study period using a generalized linear mixed model with a logit link that includes an indicator for study arm and random effects for clinic and primary care provider to account for the multilevel data structure.
Implementation quality (Aim 3a) | Up to 3 years
  The Investigators will assess implementation quality and outcomes through stakeholder interviews (patients, providers, administrators) and chart reviews. The information gained will guide adaptations of the intervention for future use so that clinicians maximize effectiveness, feasibility, acceptability, sustainability, and impact. Findings will also determine the resources needed to successfully scale the intervention to different settings
Cost effectiveness (Aim 3b) | Up to 3 years
  Will use standard cost-effectiveness techniques (including time discounting) to conduct an incremental cost-effectiveness analysis, measuring the Incremental Cost-Effectiveness Ratio of the natural language processing-based electronic health record intervention compared to usual care office outreach.

SECONDARY OUTCOMES:
Time from high risk neoplasia (HRN) diagnosis to colonoscopy (Aim 2) | From HRN diagnosis to colonoscopy, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Folasade P May, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] May FP, McEwan JA, Tuan JJ, Crespi CM, Maehara CK, Yang JO, Uy A, Gupta S, Kang Y, Myint A, Naini BV, Elmore JG, Kadiyala S, Ong MK, Bui AAT, Hamilton AB, Chang LC, Gelvezon A, Hsu W, Bastani R. Increasing timely colonoscopy surveillance for patients with high-risk colorectal polyps: Protocol for a cluster randomized trial. Contemp Clin Trials. 2026 Jan;160:108147. doi: 10.1016/j.cct.2025.108147. Epub 2025 Nov 17. PMID 41260460